CLINICAL TRIAL: NCT03401957
Title: A Non-interventional Uncontrolled Multicenter Study to Investigate the Emergence of RAS Resistance Mutations in RAS Wild Type mCRC Patients Receiving First Line Cetuximab Treatment
Brief Title: The Emergence of RAS Mutations in Metastatic Colorectal Cancer Patients Receiving Cetuximab Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: National Cheng-Kung University Hospital (Other); Kaohsiung Medical University Chung-Ho Memorial Hospital (Other); Taipei Veterans General Hospital, Taiwan (Other Government); Cathay General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: EC1060904
Record Dates: First submitted 2018-01-10; First posted 2018-01-17 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Colorectal Cancer; Drug Resistance; Mass Spectrometry; RAS-RAF Pathway Deregulation
Keywords: colorectal cancer; cetuximab resistance; liquid biopsy; RAS mutation
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; Liquid Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RAS wild-type colorectal cancer: RAS mutation of patients who are pathologically diagnosed as metastatic colorectal cancer with RAS wild type genotyping will be evaluated using liquid biopsy during cetuximab treatment.
  Interventions: Drug: Cetuximab; Diagnostic Test: liquid biopsy

INTERVENTIONS:
Drug: Cetuximab — Cetuximab-based infusional 5-FU regimen as the 1st line treatment.
  Other Names: erbitux
Diagnostic Test: liquid biopsy — The blood samples taken from subjects will be evaluated for RAS genotype using MassARRAY technique.

SUMMARY:
To evaluate the emergence of RAS mutation in patients with metastatic colorectal cancer, circulating free DNA will be analyzed using mass spectrometric genotyping in subjects during cetuximab treatment. The hypothesis of this study is that acquired RAS mutation is responsible for the resistance to cetuximab treatment in wild-type colorectal cancer. The usefulness of liquid biopsy to monitor dynamic genetic alterations in colorectal cancer during treatment will also be investigated in this study.

DETAILED DESCRIPTION:
This is a single arm, non-interventional, uncontrolled, multicenter study in metastatic colorectal cancer patients receiving cetuximab-based infusional 5-FU regimen as 1st line treatment. Patients who are pathologically diagnosed as metastatic colorectal cancer with RAS wild type genotyping will be recruited in this study. Patients enrolled will be those for whom it is planned to treat their colorectal cancer with a cetuximab-based infusional 5-FU regimen according to the locally approved label. Cetuximab-based treatment is anticipated to be continued until disease progression, intolerable toxic effects, or withdrawal of consent occurs. Blood samples from patients enrolled in this study will be collected before the start of cetuximab-based chemotherapy, and every 3 months during the 1st line treatment with the cetuximab-based regimen. Blood sampling is also required at 2-3 weeks after disease progression following cetuximab treatment and after disease progression on 2nd line treatment. The blood samples will be sent to a central laboratory at the Taipei Institute of Pathology and evaluated for RAS genotype, using MassARRAY technique. The objectives of this study are described as follows.

Primary objective:

To observe the percentage of detected RAS mutations (circulating DNA) during 1st line cetuximab exposure in Taiwanese patients.

Secondary objective:

1. To observe the time to onset of detected RAS mutation in circulating DNA.
2. To observe the quantification mutation load change under treatment.
3. To evaluate clinical response and resection rate of metastases with 1st line cetuximab exposure.
4. To evaluate treatment duration with 1st line cetuximab.
5. To investigate the correlation between the occurrence and levels of acquired RAS mutations post-cetuximab treatment and clinical outcomes (progression free survival and overall survival).
6. To calculate total 1st line cetuximab exposure dosage.
7. To investigate correlation between the irinotecan or oxaliplatin dosage and acquired resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically proven metastatic colorectal cancer for whom treatment with cetuximab in 1st line setting, is planned as part of routine clinical practice, as per the locally approved label and the best scientific information; the decision to prescribe cetuximab is at the sole discretion of the investigator. The choice of standard chemotherapy regimen for 1st line treatment of colorectal cancer is also at the sole discretion of the Investigator, based upon routine clinical practice.
2. Patients aged 20 years and above.
3. Patients who are molecularly diagnosed as having RAS wild-type mCRC.
4. Patients who are willing to provide blood samples during the study
5. Patients who are willing, and able and give, signed informed consent.

Exclusion Criteria:

1. Patients having a history of prior exposure to any anti-EGFR therapy.
2. Contra-indications to cetuximab as per locally approved label.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with RAS wild-type metastatic colorectal cancer receiving cetuximab-based regimen (5-FU containing) as the 1st line treatment.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of detected circulating DNA RAS mutations during 1st line cetuximab exposure. | 9 months
  Percentage of detected RAS mutations during cetuximab treatment.

SECONDARY OUTCOMES:
Time to onset of newly detected circulating DNA RAS mutation. | 9 months
  Time duration between the start of cetuximab treatment and newly detection of RAS mutation.
Mutation load (percentage of detected mutated alleles) until disease progression. | 9 months
  Percentage of detected mutated alleles at disease progression.
Percentage of detected RAS mutations at the time of progression. | 9 months
  Percentage of detected RAS mutations at the time of progression.
Clinical response rate by the investigator's judgement based on RECIST criteria. | 9 months
  Response rate of tumor after cetuximab treatment.
Resection rate of liver or lung metastases. | 9 months
  Resection rates of metastases after cetuximab treatment.
Duration of treatment with cetuximab in 1st line treatment. | 9 months
  Time duration of cetuximab as the 1st line treatment.
Total accumulated dosage of cetuximab in 1st line treatment. | 9 months
  Total accumulated dosage of cetuximab in 1st line treatment.
Progression-free survival from start of 1st line treatment with cetuximab. | 9 months
  The time duration of subjects between the inclusion in the study and disease progression.
Overall survival from the start of 1st line treatment with cetuximab. | 24 months
  The time duration of subjects between the inclusion in the study and death.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Tzong Chen, M.D., Principal Investigator — National Institute of Cancer Research, National Health Research Institutes
Locations (4):
- Taiwan (4):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - Cathay General Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

REFERENCES:
- [Derived] Tsai HL, Lin CC, Sung YC, Chen SH, Chen LT, Jiang JK, Wang JY. The emergence of RAS mutations in patients with RAS wild-type mCRC receiving cetuximab as first-line treatment: a noninterventional, uncontrolled multicenter study. Br J Cancer. 2023 Oct;129(6):947-955. doi: 10.1038/s41416-023-02366-z. Epub 2023 Jul 24. PMID 37488448
- [Derived] Chen SH, Tsai HL, Jiang JK, Sung YC, Huang CW, Yeh YM, Chen LT, Wang JY. Emergence of RAS mutations in patients with metastatic colorectal cancer receiving cetuximab-based treatment: a study protocol. BMC Cancer. 2019 Jun 28;19(1):640. doi: 10.1186/s12885-019-5826-7. PMID 31253124